CLINICAL TRIAL: NCT06414941
Title: Dexmedetomidine Combined With Esketamine Effects the Quality of Sleep
Brief Title: The Effect of Dexmedetomidine and Esketamine Combined Infusion Quality of Sleep Undergoing Modified Radical Mastectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anqing Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: errtg555
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Dexmedetomidine Plus Esketamine Affect Postoperative Sleep Quality
Keywords: Esketamine; Sleep quality; Dexmedetomidine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine on sleep quality with radical mastectomy (Experimental): Dexmedetomidine infusion Patients received dexmedetomidine (0.5 µg/kg over 10 min before the induction of anesthesia), and then dexmedetomidine was infused at a rate of 0.4 μg/kg/h until 20 min before the end of operation
  Interventions: Drug: Dexmedetomidine administration; Drug: Dexmedetomidine plus low-dose esketamine administration; Drug: Dexmedetomidine plus high-dose esketamine administration
- Dexmedetomidine plus low-dose esketamine on sleep quality with radical mastectomy (Experimental): Dexmedetomidine and low-dose eskeamine combined infusion Patients received a bolus infusion of dexmedetomidine (0.5 µg/kg) and esketamine (0.5 mg/kg)over 10 min before the induction of anesthesia, and then dexmedetomidine were infused at a rate of 0.4 µg/kg/h and 2 µg/kg/min until 20 min before the end of operation, respectively.
  Interventions: Drug: Dexmedetomidine administration; Drug: Dexmedetomidine plus low-dose esketamine administration; Drug: Dexmedetomidine plus high-dose esketamine administration
- Dexmedetomidine plus high- dose esketamine on sleep quality with radical mastectomy (Experimental): Dexmedetomidine and high-dose eskeamine combined infusion Patients received a bolus infusion of dexmedetomidine (0.5 µg/kg) and esketamine (0.5 mg/kg)over 10 min before the induction of anesthesia, and then dexmedetomidine were infused at a rate of 0.4 µg/kg/h and 4 µg/kg/min until 20 min before the end of operation, respectively.
  Interventions: Drug: Dexmedetomidine administration; Drug: Dexmedetomidine plus low-dose esketamine administration; Drug: Dexmedetomidine plus high-dose esketamine administration

INTERVENTIONS:
Drug: Dexmedetomidine administration — atients received dexmedetomidine (0.5 µg/kg over 10 min before the induction of anesthesia), and then dexmedetomidine was infused at a rate of 0.4 μg/kg/h until 20 min before the end of operation
Drug: Dexmedetomidine plus low-dose esketamine administration — Patients received a bolus infusion of dexmedetomidine (0.5 µg/kg) and esketamine (0.5 mg/kg)over 10 min before the induction of anesthesia, and then dexmedetomidine were infused at a rate of 0.4 µg/kg/h and 2 µg/kg/min until 20 min before the end of operation, respectively.
Drug: Dexmedetomidine plus high-dose esketamine administration — Patients received a bolus infusion of dexmedetomidine (0.5 µg/kg) and esketamine (0.5 mg/kg)over 10 min before the induction of anesthesia, and then dexmedetomidine were infused at a rate of 0.4 µg/kg/h and 4 µg/kg/min until 20 min before the end of operation, respectively.

SUMMARY:
BACKGROUND: Some studies have revealed that intravenous dexmedetomidine and esketamine improve the quality of sleep after surgery. The investigators investigated whether co-administration dexmedetomidine and esketamine could better improve the the quality of sleep after modified radical mastectomy.

METHODS: One hundred and five women with elective modified radical mastectomy were randomly divided into 3 groups: Patients in group D received dexmedetomidine (0.5 µg/kg over 10 min before the induction of anesthesia), and then dexmedetomidine was infused at a rate of 0.4 μg/kg/h until 20 min before the end of operation. Patients in group DE1 received a bolus infusion of dexmedetomidine (0.5 µg/kg) and esketamine (0.5 mg/kg)over 10 min before the induction of anesthesia, and then dexmedetomidine were infused at a rate of 0.4 µg/kg/h and 2 µg/kg/min until 20 min before the end of operation, respectively. Patients in group DE2 received received a bolus infusion of dexmedetomidine (0.5 µg/kg) and esketamine (0.5 mg/kg)over 10 min before the induction of anesthesia, and then dexmedetomidine were infused at a rate of 0.4 µg/kg/h and 4 µg/kg/min until 20 min before the end of operation, respectively. Primary outcome was the quality of sleep (PSQI) at the day after surgery and 1 day after surgery. The secondary outcomes included MAP, HR, postoperative VAS pain scores, side effects such as the incidence of postoperative nausea and vomiting, hallucination, as well as agitation, drowness, postoperative rescue analgesics and anti-emetics, recovery time, and extubation time.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status Ⅰ- Ⅱ
* Scheduled for elective modified radical mastectomy

Exclusion Criteria:

* Severe respiratory disease
* Renal or hepatic insufficiency
* History of preoperative psychiatric
* Preoperative bradycardia
* Preoperative atrioventricular block
* Preoperative hypertension
* BMI>30

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index (PSQI) | the day after surgery
  Our primary outcome was Pittsburgh sleep quality index (PSQI) at the day after surgery

SECONDARY OUTCOMES:
Pittsburgh sleep quality index (PSQI) | 1 day after surgery
  Our primary outcome was Pittsburgh sleep quality index (PSQI) on 1 day after surgery
pain visual analogue scale scores | The first 48 hours after operation
  Our primary outcome was pain visual analogue scale scores

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anqing Hospital Anesthesiology, Anqing, Anhui, China